CLINICAL TRIAL: NCT04679051
Title: Effect of Pulsatile Pressure and Long Sleep Duration on Cerebral Vascular Function
Brief Title: Long Sleep Duration and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Joaquin U Gonzales, PhD, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19IPLOI34760579
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Sleep
Keywords: sleep duration; blood pressure; vasodilation; cognitive function
MeSH Terms: conditions — Aneurysm | interventions — Sleep Duration

STUDY DESIGN:
Intervention Model Description: This project will be a randomized crossover study. Each week will consist of a different time in bed schedule of either 8 or 11 hours time in bed (TIB). The investigators estimated that about 11 hours in bed will result in at least 9 hours of total sleep time (i.e., long duration sleep). Laboratory testing will occur after five consecutive nights of either 8h or 11h TIB to assess the effect of sleep duration on vascular function, and after the sixth consecutive night of TIB to assess the effect of exercise on vascular function under different sleep conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 hours time in bed (Experimental): Participants will be asked to spend 8 hours time in bed with the aim of achieving one week of normal sleep duration (7 to 8 hours).
  Interventions: Behavioral: Sleep duration
- 11 hours time in bed (Experimental): Participants will be asked to spend 11 hours time in bed with the aim of achieving one week of long duration sleep as defined as 9+ hours of sleep.
  Interventions: Behavioral: Sleep duration

INTERVENTIONS:
Behavioral: Sleep duration — Participants will be asked to alter time in bed to achieve specified sleep durations.

SUMMARY:
Sleep duration has received much attention in recent years due to strong evidence that not enough sleep can increase risk for a number of diseases and disorders. Research is emerging that too much sleep also has a negative impact on health, particularly higher risk for myocardial infarction and stroke. The investigators hypothesize that long duration sleep has the ability to impair peripheral and cerebral vascular function in middle-aged to older adults.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of long duration sleep (>9 hours) to recommended levels of sleep (7-8 hours) in a crossover designed study requiring adults to maintain each prescribed sleep duration for one week. Ambulatory brachial and central aortic blood pressure will be measured during sleep, while cerebrovascular reactivity, carotid artery hemodynamics (e.g., flow pulsatility), aortic pulse wave reflections, cognitive function, and peripheral vasodilatory function will be measured before and after each sleep protocol. A secondary objective of this study is to understand whether aerobic exercise can improve vascular function under conditions of different sleep durations. This information will shed light upon the impact of sleep parameters on exercise-induced improvements in vascular function.

ELIGIBILITY:
Inclusion Criteria:

* recreationally active
* reporting no recent history of sleep problems
* not taking sleep-inducing medication
* not diabetic (fasting blood glucose <126 mg/dL)

Exclusion Criteria:

* show symptoms of insomnia
* smoke
* have a personal history of stroke or diabetes
* take birth control pills

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin U Gonzales, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected or generated from the project will be made available on ClinicalTrials.gov within 12 months from the primary completion date
Supporting Information: ICF
Time Frame: All data collected or generated from the project will be made available on ClinicalTrials.gov within 12 months from the primary completion date.
Access Criteria: Open access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 participants were screened for eligibility between October 16, 2019 and May 24, 2021at Texas Tech University in Lubbock, TX.
Pre-assignment Details: 23 of 34 participants were randomized. Of those not randomized, 8 did not meet inclusion criteria and 3 declined to participate.
Groups:
- 8, Then 11 Hours in Bed: Participants were first asked to spend 8 hours in bed for one week. After 1 night of washout, participants were then asked to spend 11 hours in bed for one week.
- 11, Then 8 Hours in Bed: Participants were first asked to spend 11 hours in bed for one week. After 1 night of washout, participants were then asked to spend 8 hours in bed for one week.
Period: Overall Study
Arm/Group | 8, Then 11 Hours in Bed | 11, Then 8 Hours in Bed
Started | 12 | 11
Completed | 6 | 6
Not Completed | 6 | 5
Not completed — felt tired after restricted time in bed | 3 | 0
Not completed — discomfort with blood pressure cuff | 2 | 0
Not completed — scheduling conflict | 1 | 1
Not completed — Protocol Violation | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8, Then 11 Hours in Bed | 11, Then 8 Hours in Bed | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (6) | 43 (3) | 45 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26 (3) | 24 (5) | 26 (4)
Seated Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 118 (10) | 111 (8) | 114 (9)
Seated Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 75 (6) | 73 (10) | 74 (8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Wake in Central Aortic Pulse Pressure After 11 Hours in Bed
Description: Central aortic pulse pressure was measured one night during the week of 8 hours in bed, then again one night during the week of 11 hours in bed. Blood pressure was measured using an Oscar2 ambulatory blood pressure device. The device started recordings one hour prior to sleep and was programmed to take measurements once every 30 minutes during sleep until 10:00pm then every 45 minutes after 10:00pm until participants arose from bed. The change in central aortic pulse pressure from being awake to being asleep was compared between 8 and 11 hours in bed conditions.
Time Frame: One night during each time in bed condition
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- 8 Hours in Bed: Condition in which participants spent 8 hours in bed for one week.
- 11hours in Bed: Condition in which participants spent 11 hours in bed for one week.
Arm/Group | 8 Hours in Bed | 11hours in Bed
Number analyzed (Participants) | 12 | 12
mm Hg | -1.5 (8.9) | 0.5 (5.2)
Statistical Analysis 1: Comparison: 8 Hours in Bed vs 11hours in Bed; Two-tailed paired t-tests were used to compare variables between time in bed conditions; Test type: Superiority; p = 0.36, t-test, 2 sided

2. Primary Outcome: Change in Cerebral Vascular Reactivity After 11 Hours in Bed
Description: Blood flow measured in the middle cerebral artery during hypercapnia was measured after one week of 8 hours in bed, then again after one week of 11 hours in bed. Cerebral blood flow was measured using transcranial Doppler during 3 minutes of transient hypercapnia induced by rebreathing. Cerebral vascular reactivity was considered as the percent increase in cerebral blood flow at the end of 3 minutes of rebreathing relative to the Torr change in end-tidal carbon dioxide (percent change/Torr).
Time Frame: Morning after one week of 8 and 11 hours in bed
Population: The middle cerebral artery could not be located in 3 participants, so data was analyzed in 9 participants that had complete data.
Measure: Mean (Standard Deviation); unit: percent change/Torr
Groups:
- 11 Hours in Bed: Condition in which participants spent 11 hours in bed for one week.
Arm/Group | 8 Hours in Bed | 11 Hours in Bed
Number analyzed (Participants) | 9 | 9
percent change/Torr | 11.9 (2.8) | 11.3 (1.8)
Statistical Analysis 1: Comparison: 8 Hours in Bed vs 11 Hours in Bed; Paired t-test comparing the two time in bed protocols; Test type: Superiority; p = 0.51, t-test, 2 sided

3. Primary Outcome: Change in Peak Reactive Hyperemia After 11 Hours in Bed
Description: Peak forearm blood flow was measured after one week of 8 hours in bed, then again after one week of 11 hours in bed. Peak reactive hyperemia in the forearm (ml/100ml/min) was measured using venous occlusion plethysmography after 10 minutes of forearm ischemia resulting from blood pressure cuff inflation at the upper-arm. Peak blood flow was considered the highest blood flow measurement after the blood pressure cuff was deflated.
Time Frame: Morning after one week of 8 and 11 hours in bed
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: ml/100ml/min
Arm/Group | 8 Hours in Bed | 11 Hours in Bed
Number analyzed (Participants) | 12 | 12
ml/100ml/min | 20.8 (5.8) | 24.2 (7.2)
Statistical Analysis 1: Comparison: 8 Hours in Bed vs 11 Hours in Bed; Paired t-test comparing peak forearm blood flow between sleep protocols; Test type: Superiority; p = 0.03, t-test, 2 sided

4. Primary Outcome: Change in Arterial Stiffness After 11 Hours in Bed
Description: Arterial stiffness was measured after one week of 8 hours in bed, then again after one week of 11 hours in bed. Carotid-femoral pulse wave velocity was used as the measure of arterial stiffness. Radial arterial tonometry was used to derive a central aortic blood pressure wave. Wave separation analysis of the aortic pressure wave was then used to calculate pulse wave velocity from transit time and carotid-femoral path length.
Time Frame: Morning after one week of 8 and 11 hours in bed
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | 8 Hours in Bed | 11 Hours in Bed
Number analyzed (Participants) | 12 | 12
m/s | 6.84 (0.64) | 6.96 (0.64)
Statistical Analysis 1: Comparison: 8 Hours in Bed vs 11 Hours in Bed; Paired t-test used to compare carotid-femoral pulse wave velocity (index of arterial stiffness) between sleep protocols; Test type: Superiority; p = 0.29, t-test, 2 sided

5. Secondary Outcome: Change in Spatial Orientation After Aerobic Exercise
Description: Score from a Manikin test of spatial orientation that participants took using a computer with automated software (Automated Neuropsychological Assessment Metrics, known as ANAM). Scores reflect "throughput scores" which is a continuous variable that is the ratio of correct answers per minute during the Manikin test. Higher throughput scores mean better outcome, in this case, better spatial orientation ability. Participants took the Manikin test after one week of 8 and 11 hours in bed (i.e., baseline) then the morning after one day of aerobic exercise. Exercise consisted of three sessions of 10 minutes brisk walking at a heart rate considered to be moderate intensity (50-70% of age-predicted maximal heart rate). Results reported reflect the change in throughput scores after exercise (morning after exercise minus baseline).
Time Frame: Baseline and after exercise
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: correct answers per minute
Arm/Group | 8 Hours in Bed | 11 Hours in Bed
Number analyzed (Participants) | 12 | 12
correct answers per minute | 7.0 (4.7) | 3.9 (5.6)
Statistical Analysis 1: Comparison: 8 Hours in Bed vs 11 Hours in Bed; A two-way repeated measures ANOVA was used to evaluate the main effect of exercise (before vs. after exercise) on Manikin throughput scores; Test type: Superiority; p < 0.001, ANOVA — Null hypothesis is that there was no difference in change of spatial ability following one day of aerobic exercise. The ANOVA test was performed with a significance level of 0.05 (two-sided)

6. Secondary Outcome: Change in Executive Function After Aerobic Exercise
Description: Executive function was assessed using a Stroop color-word test that participants took using a computer with automated software (Automated Neuropsychological Assessment Metrics, known as ANAM). Score reported are number of correct answers. A higher score means a better outcome, in this case, better executive functioning. Participants took the Stoop color-word test after one week of 8 and 11 hours in bed (i.e., baseline) then the morning after one day of aerobic exercise. Exercise consisted of three sessions of 10 minutes brisk walking at a heart rate considered to be moderate intensity (50-70% of age-predicted maximal heart rate). Results reported reflect the change in score after exercise (morning after exercise minus baseline).
Time Frame: Baseline and after exercise
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: correct answers
Groups:
- 8 Hours Time in Bed: Change in cognitive variable following exercise within 8 hour time in bed protocol
- 11 Hours Time in Bed: Change in cognitive variable following exercise within 11 hour time in bed protocol
Arm/Group | 8 Hours Time in Bed | 11 Hours Time in Bed
Number analyzed (Participants) | 12 | 12
correct answers | 4.5 (5.4) | 2.4 (6.8)
Statistical Analysis 1: Comparison: 8 Hours Time in Bed vs 11 Hours Time in Bed; A two-way repeated measures ANOVA was used to evaluate the main effect of exercise (before vs. after exercise) on the number of correct answers during a Stroop color-word test; Test type: Superiority; p = 0.04, ANOVA — Null hypothesis is that there was no difference in the change of executive function following one day of aerobic exercise. The ANOVA test was performed with a significance level of 0.05 (two-sided)

7. Secondary Outcome: Change in Mental Flexibility After Aerobic Exercise
Description: Mental flexibility was assessed using a Switching task that participants took on a computer with automated software (Automated Neuropsychological Assessment Metrics, known as ANAM). Scores reflect "throughput scores" which is a continuous variable that is the ratio of correct answers per minute during the Manikin test. Higher throughput scores mean better outcome, in this case, better mental flexibility. Participants took the Switching task after one week of 8 and 11 hours in bed (i.e., baseline) then the morning after one day of aerobic exercise. Exercise consisted of three sessions of 10 minutes brisk walking at a heart rate considered to be moderate intensity (50-70% of age-predicted maximal heart rate). Results reported reflect the change in throughput scores after exercise (morning after exercise minus baseline).
Time Frame: Baseline and after exercise
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: correct answers per minute
Arm/Group | 8 Hours in Bed | 11 Hours in Bed
Number analyzed (Participants) | 12 | 12
correct answers per minute | 2.8 (4.9) | 1.6 (3.3)
Statistical Analysis 1: Comparison: 8 Hours in Bed vs 11 Hours in Bed; A two-way repeated measures ANOVA was used to evaluate the main effect of exercise (before vs. after exercise) on throughput scores from a Switching task; Test type: Superiority; p = 0.02, ANOVA — [p-value comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: One week for each intervention (time in bed protocol).
Description: Population included all participants who started the study.
Groups:
- 8 Hours in Bed: Participants were first asked to spend 8 hours in bed for one week. After 1 night of washout, participants were then asked to spend 11 hours in bed for one week.
- 11 Hours in Bed: Participants were first asked to spend 11 hours in bed for one week. After 1 night of washout, participants were then asked to spend 8 hours in bed for one week.
Arm/Group | 8 Hours in Bed | 11 Hours in Bed
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT04679051/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04679051/ICF_000.pdf